CLINICAL TRIAL: NCT05646537
Title: Effect of Neuro-Linguistic Programming on Comfort Level After Cesarean: A Randomized Controlled Trial
Brief Title: Cesarean Neuro Linguistic Programming Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toros University (Other)
Responsible Party: Principal Investigator, Aysel DOĞAN, Assist. Prof., Toros University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: TorosUn
Record Dates: First submitted 2022-11-10; First posted 2022-12-12 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Cesarean Section Complications
Keywords: Nurse; NLP; pain; Cesarean; nonpharmacological; holistic care; postpartum; perianesthesia process; surgery
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: NLP techniques will be applied to the experimental group, and no intervention will be applied to the control group.
Who Masked: Participant
Masking Description: Participants will not know they are in the experimental or control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The group to which NLP techniques will be applied (Experimental): After the participant consented to participate in the study with the Informed Consent Form, her comfort level was measured with the Postpartum Comfort Scale.
  A session of NLP (30 minutes) was applied to the participant. The patient was informed about the application. The mother was asked to sit or lie down i Before the discharge of the participant from the hospital, her comfort level was evaluated once again by using the Postpartum Comfort Scale
  Interventions: Behavioral: Neuro-Linguistic Programming Techniques
- Control group (No Intervention): After the participant consented to participate in the study with the Informed Consent Form, her comfort level was measured with the Postpartum Comfort Scale.
  Without having any additional practice, the participant solely had the routine clinical protocol.
  Before the discharge of the participant from the hospital, her comfort level was evaluated once again by using the Postpartum Comfort Scale.

INTERVENTIONS:
Behavioral: Neuro-Linguistic Programming Techniques — The new behavior creation technique of NLP is based on the argument that the imagination process and reality are recorded in the same way in the brain.
  Using the Participant's eye movements and imagination . He will be asked to imagine himself while caring for the stoma. participient will then be asked to re-enact the process with the correct stages of stoma care and the jurals that must be adhered to in order to successfully care for it.
  Questions will be asked about where he can find the support he needs to carry out this process successfully. At the end of this whole process, he will be expected to construct what life is like with a stoma.The technique will be applied to the patient once and will be instructed to remember this successful process every time he or she feels distressed about the stoma.
  At the end of 6 months, the quality of life and compliance will be evaluated by asking the scale questions again.
  Arms: The group to which NLP techniques will be applied

SUMMARY:
The aim of this study is to examine the effect of NLP techniques on stoma compliance and quality of life in patients with stoma.

The study will be conducted using a prospective randomized controlled single-blind clinical trial model.

The research will consist of patients with temporary or permanent colostomy/ileostomy, who are hospitalized in Mersin City Training and Research Hospital.

Research data will be obtained with demographic questionnaire, Adjustment Scale for Individuals with Ostomy and Stoma Quality of Life Scale.

Analysis of the study data will be done through the IBM SPSS Statistics 26 package program. While evaluating the study data, frequencies (number, percentage) for categorical variables and descriptive statistics (mean, standard deviation) for numerical variables will be given.

Statistical significance in the analyzes will be interpreted at the 0.05 level.

DETAILED DESCRIPTION:
Stomas are formed in order to provide stool output after surgery in cases that require removal of the bowel due to disease or trauma (Harputlu & Özsoy, 2016). Stoma surgery is a vital surgical intervention. However, the individual may have to cope with many problems that may negatively affect the adaptation process and quality of life in terms of living with a stoma. The literature is that despite the developing stoma products and professional nurse educators, the problems related to stoma compliance and quality of life of the patients continue, and complications affecting coping with these processes are seen at different rates.

The aim of this study is to examine the effect of NLP techniques on stoma compliance and quality of life in patients with stoma.

The study will be conducted using a prospective randomized controlled single-blind clinical trial model.

The study will consist of patients with temporary or permanent colostomy/ileostomy, who are hospitalized in Mersin City Training and Research Hospital.

Research data will be obtained with demographic questionnaire, Adjustment Scale for Individuals with Ostomy and Stoma Quality of Life Scale.

Analysis of the study data will be done through the IBM SPSS Statistics 26 package program. While evaluating the study data, frequencies (number, percentage) for categorical variables and descriptive statistics (mean, standard deviation) for numerical variables will be given.

The normality assumptions of the numerical variables according to the groups were examined with the Kolmogorov Smirnov test of normality and it was observed that the variables were normally distributed. For this reason, parametric statistical methods will be used in the study.

Relationships between two independent categorical variables were interpreted by Chi-square analysis. The differences between the two independent groups were examined using the Independent Sample T Test. The differences between the two dependent numerical variables will be examined with Dependent Sample T. Statistical significance in the analyzes will be interpreted at the 0.05 level.

ELIGIBILITY:
Inclusion Criteria:

* Having a c-section for the first time, being within the period after a minimum of 6 hours and before a maximum of 24 hours following the c-section,
* agreeing to participate in the study,
* not using patient-controlled analgesics, not having an additional health problem, except the c-section incision, which will likely lead to pain in the postpartum period,
* speaking and understanding Turkish, having no disability limiting mobility

Exclusion criteria:

* Mothers who wanted to withdraw from the research in any stage after being included in the sample,
* who could not have verbal communication,
* who had a hearing or visual problem, and who were previously diagnosed with a psychiatric disease were excluded from the research sample.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — woman
Enrollment: 100 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
stoma compliance scores of the participants | 1th day
  At the end of the firsth day to measure the comfort level of the participants, the average score of the Individual with a postpartum comfort Scale will be calculated The General Comfort Questionnaire developed by Kolcaba (1992). Designed as a five-point Likert-type scale, the PCS has 34 items. In this respect, the participants respond to PCS items by rating them from 1 point to 5 points. In positively worded items, "I strongly agree" refers to the highest level of comfort whilst "I strongly disagree" points to the lowest level of comfort. Negatively worded items were reverse-coded. The minimum and maximum scores to be obtained from the PCS are successively 34 and 170 points. There is no cut-off point for the PCS. As the scores obtained from the PCS increase, the comfort levels also go up. Cronbach's alpha coefficient as the measure of internal consistency was found as 0.78 for the PCS

SECONDARY OUTCOMES:
comfort level of the participants | 3th day
  At the end of the 3th day to measure the comfort level of the participants, the average score of the Individual with a postpartum comfort Scale will be calculated The General Comfort Questionnaire developed by Kolcaba (1992). Designed as a five-point Likert-type scale, the PCS has 34 items. In this respect, the participants respond to PCS items by rating them from 1 point to 5 points. In positively worded items, "I strongly agree" refers to the highest level of comfort whilst "I strongly disagree" points to the lowest level of comfort. Negatively worded items were reverse-coded. The minimum and maximum scores to be obtained from the PCS are successively 34 and 170 points. There is no cut-off point for the PCS. As the scores obtained from the PCS increase, the comfort levels also go up. Cronbach's alpha coefficient as the measure of internal consistency was found as 0.78 for the PCS

CONTACTS AND LOCATIONS:
Locations (1):
- Toros University, Mersin, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
One year after the study results were published in a scientific journal
Supporting Information: Study Protocol, CSR
Time Frame: 48th months
Access Criteria: With the permission of the principal investigator

REFERENCES:
- [Derived] Dogan A, Dal NA, Beydag KD. Effect of neuro-linguistic programming on comfort after cesarean: a randomized controlled trial neuro-linguistic programming comfort level cesarean. BMC Pregnancy Childbirth. 2025 Aug 30;25(1):902. doi: 10.1186/s12884-025-08043-8. PMID 40885918